CLINICAL TRIAL: NCT07107139
Title: Influence of Authorized Smokeless Tobacco Product Modified Risk Claims II: Laboratory Assessment of Sensory and Subjective Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: I-4008824-1; R21CA289541 (NIH)
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Smokeless Tobacco
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Copenhagen group (Active Comparator): Participants will place .66 grams of Copenhagen between cheek and gums for up to 30 minutes.
  Interventions: Other: Copenhagen group
- Snus Group (Active Comparator): Participants will place one pouch of snus beween cheek and gums for up to 30 minutes.
  Interventions: Other: Snus group

INTERVENTIONS:
Other: Copenhagen group — Participants use product for up to 30 minutes
  Arms: Copenhagen group
Other: Snus group — Participants use product for up to 30 minutes
  Arms: Snus Group

SUMMARY:
This study seeks to measure the effects of smokeless tobacco product risk messages on sensory experiences and future intentions to use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years of age
* Residing in 8 counties of Western NY (Erie, Niagara, Cattaraugus, Chautauqua, Allegheny, Livingston, Genesee, Orleans, Wyoming)
* Smoke cigarettes every day, at least 5 cigarettes per day, for at least 1 year
* Open to trying a non-combusted oral tobacco product
* Have the ability to read, write, and communicate in English
* Have successfully completed our preliminary Auction study I-4008824 with a bid for Copenhagen and/or General Snus > $0
* Willing to abstain smoking 8-10 hours prior to each laboratory session and complete breath CO test for verification (<8ppm)
* Female participants must be amenable to taking a pregnancy test (urine) prior to beginning study procedures.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Age ≥ 21 years of age
* Residing in 8 counties of Western NY (Erie, Niagara, Cattaraugus, Chautauqua, Allegheny, Livingston, Genesee, Orleans, Wyoming)
* Smoke cigarettes every day, at least 5 cigarettes per day, for at least 1 year
* Open to trying a non-combusted oral tobacco product
* Have the ability to read, write, and communicate in English
* Have successfully completed our preliminary Auction study I-4008824 with a bid for Copenhagen and/or General Snus > $0
* Willing to abstain smoking 8-10 hours prior to each laboratory session and complete breath CO test for verification (<8ppm) .
* Female participants must be amenable to taking a pregnancy test (urine) prior to beginning study procedures.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in sensory response | Before viewing study ads and immediatley after viewing
  assessed with a 0-100 visual analog scale - anchored by word descriptors at each end.

SECONDARY OUTCOMES:
Change in nicotine boost | Will be collected after 5, 15 and 30 minutes of product use.
  Will be measured after use of products with gas chromatography-mass spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Roswell Park, Buffalo, New York, United States